CLINICAL TRIAL: NCT06417645
Title: the BIS Index Response is Poorly Described by Propofol Effect Site Eleveld's Model After Applying a Perturbation
Brief Title: Re-evaluation of the Effect Site Model of the PKPD Propofol Eleveld Model
Acronym: Eleved PD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Pablo O. Sepulveda, Dr. Med, Universidad del Desarrollo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEC-SSLR ord: 459
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy; Surgery
Keywords: propofol, Eleveld, BIS, predicted effect site model, non-lineal behavior

STUDY DESIGN:
Intervention Model Description: healthy patients proposed for elective surgery longer than 60 min, received a standard protocol TCI iv anesthesia with EEG BIS index monitoring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIS predicted vs real (Experimental): After slow propofol induction and standard monitoring with BIS EEG monitor. The propofol infusion guided by iTIVA simulator (Android / iOS) using Eleveld kinetic model. LOC (defined as loss of response to loud call and shoulder movement-touch), the same concentration of propofol will be maintained for 5 minutes to assess EEG stability. .Intubation will proceed as usual, starting remifentanil at 4.5 ng/ml and rocuronium bromide 0.6 mg/kg. After 5 min and before the start of surgery, propofol will be infused at 15 mg/kg/h until 1% BSR is reached, observed on the BIS monitor, and then return to the rate that represents the LOC concentration. EEG data shall be retrieved from the BIS monitor via USB. Post hoc using the software tivatrainer.com we will simulate the Eleved calculated plasma concentration and the Bis prediction with our BIS real data.
  Interventions: Drug: fixed propofol infusion 15 mg/kg/h until 1% BSR (burst suppression ratio)

INTERVENTIONS:
Drug: fixed propofol infusion 15 mg/kg/h until 1% BSR (burst suppression ratio) — after a slow induction with propofol to loss of consiousness (LOC), we proceed to give remifentanil TCI and rocuronium and intubate the patient. After 5 min we infuse 15 mg/kg/h until 1%BSR observe in the BIS monitor. Then we reduce the TCI LOC predicted concentration.

SUMMARY:
in healthy patients undergoing elective surgery, after a very slow induction, using Eleveld's kinetics as a reference, after loss of consciousness (LOC) and intubation, proceed to infuse propofol until 1% burst suppression ratio is obtained. Then return to the LOC concentration. The BISindex predicted by the model and the real one will be evaluated. The evolution of spectral density frequencies over time will also be evaluated.

DETAILED DESCRIPTION:
Eleveld is a recently developed PKPD model of propofol, which includes multiple covariates in its pharmacokinetics.

This model, called Universal, includes data from all studies conducted with plasma levels in the world, where the principal investigator (PSV) has been directly involved.

For pharmacodynamics (PD), Eleveld, includes processed electroencephalogram (EEG) readings, but only by nominal BIS index.

The use of BIS as a unique marker of propofol hypnosis shows multiple limitations as it results from a computer algorithmic application, which can be influenced by drugs, inter-individual variability, among others.

Therefore, to determine the effect there are nowadays more accurate tools such as spectrogram processing and determination of alpha power by spectral density (PDS).

This project aims to re-evaluate the modelling of the temporal behaviour of the effect in the BIS index, using the reference of the Eleveld kinetic model, associated to a spectrogram that allows the evaluation of the alpha and delta band dynamics as a predictor of the propofol effect.

In our study we intend to replace the BIS value by the alpha and delta power progress in decibels (dB) and eventually build a pharmacodynamic (PD) model with a marker more associated to the specific cortical electrical phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients between 18 and 60 years of age, who undergo elective surgery in the central ward of the Hospital Base San José Osorno, Chile. Consecutive patients from the beginning of the study up to 12 months from the admission of the first patient.

Exclusion Criteria:

* Emergency surgery patient.
* Patients with dementia, delirium or altered state of consciousness.
* Full stomach or risk of aspiration.
* Allergic to propofol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-09-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
predicted BIS index vs real BIS index | anesthesia
  we compare the BIS predicted from the Eleveld model vs the response of our patients uring all the anesthesia procedure

SECONDARY OUTCOMES:
evaluation of the evolution of the EEG frequency bands | anesthesia
  Evaluate the differents EEG frequency bands at LOC, at maximal perturbation and when we reach again the LOC predicted concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Base san José de Osorno, Osorno, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sepulveda PO, Mora X. [Reevaluation of the time course of the effect of propofol described with the Schnider pharmacokinetic model]. Rev Esp Anestesiol Reanim. 2012 Dec;59(10):542-8. doi: 10.1016/j.redar.2012.07.019. Epub 2012 Oct 4. Spanish. PMID 23040653
- [Result] Eleveld DJ, Colin P, Absalom AR, Struys MMRF. Pharmacokinetic-pharmacodynamic model for propofol for broad application in anaesthesia and sedation. Br J Anaesth. 2018 May;120(5):942-959. doi: 10.1016/j.bja.2018.01.018. Epub 2018 Mar 12. PMID 29661412